CLINICAL TRIAL: NCT01109823
Title: Pharmacokinetic Evaluation of Fluoroquinolone Antibiotics Administered Intravenously in Intensive Care Patients With Normal Renal Function and With Renal Hyperfiltration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/167
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Infection
Keywords: Patients hospitalized at Intensive Care Unit treated with levofloxacin IV
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with normal renal function (Active Comparator): Patients with normal renal function hospitalized at the Department Intensive Care Unit who are being treated with levofloxacin I.V. (500mg, twice daily) for an infection.
  Interventions: Drug: intravenous administration of levofloxacin
- patients with hyperfiltration (Active Comparator): Patients with hyperfiltration hospitalized at the Department Intensive Care Unit who are being treated with levofloxacin I.V. (500mg, twice daily) for an infection.
  Interventions: Drug: intravenous administration of levofloxacin

INTERVENTIONS:
Drug: intravenous administration of levofloxacin — Intravenous administration of levofloxacin is used.

SUMMARY:
At the intensive care unit (ICU) fluoroquinolone antibiotics, like levofloxacin, are frequently used for the treatment of infections.

Adequate blood levels are required for a good efficacy of the antibiotic. Due to the fact that levofloxacin is almost completely eliminated renally, the blood levels for this antibiotic are strongly influenced by the renal function. Therefore, this study aims to evaluate the pharmacokinetics of levofloxacin in patients with hyperfiltration, in comparison with critically ill patients with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at the Department Intensive Care Unit who are being treated with levofloxacin I.V. (500mg, twice daily) for an infection.

Exclusion Criteria:

* Younger than 18 years
* No informed consent
* No arterial catheter
* Hematocrit ≤ 21
* Pregnancy and lactation
* Creatinine clearance < 80 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the pharmacokinetics of levofloxacin in patients with hyperfiltration, in comparison with critically ill patients with normal renal function. | 12 hours after start antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Bocxlaer, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - University Ghent, Ghent
  - University Hospital Ghent, Ghent